CLINICAL TRIAL: NCT00520156
Title: Analysis of the Prevalence and Characteristics of Co-Morbid Sleep and Headache Disorders in Patients Being Evaluated at the WRAMC Sleep Disorders Laboratory, and the Efficacy of CPAP Treatment on Headache Burden in Obstructive Sleep Apnea Patients With a Co-Morbid Headache Disorder
Brief Title: Analysis of the Prevalence and Characteristics of Concomitant Sleep and Headache Disorders, and the Efficacy of CPAP Treatment for Headache Among Those Patients Diagnosed With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: 07-17021
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Headache Disorder; Sleep Disorder; Obstructive Sleep Apnea
MeSH Terms: conditions — Headache Disorders; Sleep Wake Disorders; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Patients diagnosed with obstructive sleep apnea (OSA) will be offered standard of care treatment of CPAP (patients given oral appliances for OSA are excluded from our study). Note: our study is a survey-based and observational study following patients who are being evaluated for sleep disorders. Those patients diagnosed with OSA would be offered CPAP or possibly an oral appliance regardless of whether they are entered into our study or not.

SUMMARY:
There is a well-documented but poorly understood relationship between headache disorders (e.g. migraine, cluster headaches, awakening headaches, etc.) and sleep disorders. One hypothesis includes an underlying disorder known as obstructive sleep apnea (OSA) with low overnight oxygen saturations and possibly elevated carbon dioxide levels which result in awakening headache. Bruxism, or grinding of the teeth, has also been anecdotally associated with headache. The converse of these arguments is that the patient may have a primary headache disorder, for example migraine, leading to disordered sleep patterns or insomnia. The true relationship between the two, as alluded above, is unknown. The actual prevalence of the two disorders occurring simultaneously is not known.

There have been several small, retrospective studies which have attempted to evaluate this relationship. One of these studies evaluated those patients diagnosed with OSA who were given the standard of care therapy - continuous positive airway pressure (CPAP) - and found that headaches among these patients were improved after using CPAP. Again, this was a small, retrospective study.

We propose a study whereby patients who are referred for polysomnography (PSG, or "sleep study") are consented, then surveyed on the presence or absence of headache. A brief questionnaire is followed up with a more detailed questionnaire to characterize whether this headache that the patient has is truly a headache disorder. Following the survey and PSG, the patient's sleep study parameters are evaluated to see whether there are certain correlations between what has been recorded and the particular headache disorder present.

Lastly, if the patient was diagnosed with OSA and fitted with a CPAP device, the patient will be queried several weeks later to evaluate whether there was improvement or cessation of the headache disorder.

DETAILED DESCRIPTION:
There is a well-documented but poorly understood relationship between headache disorders (e.g. migraine, cluster headaches, awakening headaches, etc.) and sleep disorders. The exact prevalence of patients with concomitant headache disorder and sleep disorder is not even known. Hypotheses surrounding the relationship include low overnight oxygen saturation and/or hypercarbia in the case of obstructive sleep apnea (OSA) with awakening headache, primary headache disorder as a contributor to secondary sleep disorder, atypical lengths or percentages of time in various sleep stages resulting in disordered sleep patterns and subsequent headache, bruxism causing tension type headaches, among others. Our review of the literature shows there has not yet been a prospective trial evaluating headache disorders and concomitant sleep disorders with attempts to find vagaries or abnormalities in terms of sleep parameters as a way to explain headache disorder.

Additionally, although there have been few retrospective reviews of small numbers of patients examining an intervention (in this case, the addition of continuous positive airway pressure - CPAP) as a means to correct a sleep disorder with a subsequent evaluation of the patient's pre-existing headache disorders, there has yet to be a prospective trial evaluating same. Our team identified at least one retrospective study that would suggest that treating OSA with standard of care CPAP improved pre-existing symptoms of headache.

Our study proposes to - after obtaining consent - survey patients with suspected sleep disorders who have been scheduled for a sleep study to evaluate the overall prevalence of headache disorder among this particular population. We would then evaluate various standard sleep study parameters such as lowest oxygen saturation, time in various sleep stages, sleep latency, total sleep time, respiratory disturbance index, presence of bruxism, and so on, to see whether there is a correlation between certain of these parameters and a particular headache disorder. We also would survey those patients diagnosed with OSA following institution of CPAP to see whether there was a decrement or cessation in headache frequency or intensity.

Being that a significant proportion of our patients are returning war veterans with possible traumatic brain injuries or post-traumatic stress disorder, we would also query patients regarding the presence of these disorders. These data would be taken into account as a sub-analysis of the overall data set.

The study will be of 12 months duration. Over 2000 sleep studies are performed at our institution in 12 months. We anticipate an enrollment of between 400 to 800 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been screened at the Walter Reed Army Medical Center (WRMAC) sleep clinic with chief complaint of sleep disorder and have been scheduled for an overnight PSG at WRAMC. Sleep symptoms may include such difficulties as initiating sleep, maintaining sleep, disturbed sleep, not feeling refreshed in the morning, sleepiness during the day, and snoring
* Ages 18-80
* Satisfactory completion of sleep and headache inventory
* Satisfactory completion of overnight polysomnogram
* May have used sleeping preparations
* May have used anti-migraine medication
* May have other medical conditions and be on other medications

Exclusion Criteria:

* Age below 18 or over 80
* Inability to understand and sign an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Quast, MD, Principal Investigator — Pulmonary, Critical Care, and Sleep Medicine; National Capital Consortium, Washington, DC
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States